CLINICAL TRIAL: NCT04276610
Title: Words on the Brain: Can Reading Rehabilitation for Age-Related Vision Impairment Improve Cognitive Functioning?
Acronym: WOTB
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID-19 has delayed the study recruitment beyond the available funding
Sponsor: Université de Montréal (Other)
Collaborators: Fonds de la Recherche en Santé du Québec (Other Government); Canadian Institutes of Health Research (CIHR) (Other Government)
Responsible Party: Principal Investigator, Walter Wittich, Assistant Professor, Université de Montréal
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CRIR-1284-1217
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2023-04-03 (Actual); Status verified 2023-03

CONDITIONS: Age-related Macular Degeneration; Dementia; Low Vision; Low Vision Aids; Hearing Loss; Reading Problem; Cognitive Impairment
MeSH Terms: conditions — Macular Degeneration; Dementia; Vision, Low; Hearing Loss; Cognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Healthy Control Participants (No Intervention): Older adults (65+) without impairments in vision or hearing. This groups will simply be followed for the study period (1 year), measured at 6 months intervals, to provide control comparison data for all outcome measures
- Low Vision Participants (Experimental): Older adults (65+) with impairments in vision but without hearing impairment. This groups will receive regular standard of low vision rehabilitation care and will be followed for the study period (1 year), measured at 6 months intervals.
  Interventions: Behavioral: Low Vision Reading Rehabilitation
- Dual Sensory Impairment Participants (Experimental): Older adults (65+) with impairments in both vision hearing hearing. This groups will receive regular standard of low vision rehabilitation care and will be followed for the study period (1 year), measured at 6 months intervals.
  Interventions: Behavioral: Low Vision Reading Rehabilitation

INTERVENTIONS:
Behavioral: Low Vision Reading Rehabilitation — Following Time 1, participants will receive the full complement of vision rehabilitation services available and deemed suitable by their clinical staff and rehabilitation professionals of either rehabilitation centre, according to the provision of assistive devices and services regulated by the Quebec Health Insurance (RAMQ). These services are include but are not limited to: a full optometric exam to determine functional vision, including refraction and the prescription of appropriate near and distance glasses and optical devices, an assessment by a low vision therapist and/or occupational therapist, the loan provision of hand-held optical magnification devices, electronic non-optical magnification devices (e.g., portable or table-top closed-circuit televisions), or computer software for screen content magnification (e.g., ZoomText), with appropriate training and follow-up sessions in the home, if required.
  Other Names: Use of magnification devices
  Arms: Dual Sensory Impairment Participants; Low Vision Participants

SUMMARY:
Age-related vision impairment and dementia both become more prevalent with increasing age. Research into the mechanisms of these conditions has proposed that some of their causes (e.g., macular degeneration/glaucoma and Alzheimer's disease) could be symptoms of an underlying common cause, or may be equally linked to a multifactorial context in frailty and aging. Research into sensory-cognitive aging has provided preliminary data that sensory decline may be linked to the progression of dementia through the concept of sensory deprivation. Preliminary data in hearing loss rehabilitation support the idea that improved hearing may have a beneficial effect on cognitive functioning; however, there are to date no data available to examine whether low vision rehabilitation, specifically for reading, could have an equally protective or beneficial effect on cognitive health. The present proposal aims to fill this gap.

DETAILED DESCRIPTION:
The research questions are the following:

1. Does low vision rehabilitation reduce reading effort?
2. If so, does reduced reading effort increase reading activity,
3. If so, does increased reading activity improve cognitive (memory) functioning?

The objectives are to:

* Evaluate cognitive functioning and memory before, and 6 and 12 months after low vision reading rehabilitation using magnification in patients with age-related macular degeneration or glaucoma, compared to age-matched visually impaired controls who undergo rehabilitation that is NOT related to reading (e.g., mobility)
* Correlate participant characteristics with all cognitive outcome variables in order to identify potential mediators, moderators or confounders

Hypotheses:

* Measures of reading (subjective and objective effort) will be statistically significantly reduced after participants have received strategies and tools to facilitate reading.
* Measures of reading behaviour will be negatively correlated with measures of reading effort (e.g., participants who report less effort will read more, more frequently and for longer)
* Individuals that demonstrate reduced reading effort/improved reading behaviour will demonstrate improved scores on cognitive tests after 6 months of having received rehabilitation strategies and tools, compared to those whose reading effort remains high or whose reading behaviour remains unchanged. These beneficial effects will be maintained after 12 months.

Methodology

Study Design: The study utilizes a quasi-experimental approach (nonrandomized, pre-post intervention study), an approach frequently used during the evaluation of health interventions. Specifically, a 2x3 design (2 groups x 3 time points) will allow for the examination of whether cognitive performance will change before and after 6 and 12 months of a low vision reading intervention, when comparing low vision patients to age-matched controls. Participants will also be audio-recorded throughout several of the tasks to not only ensure the highest level of precision when inputting and analyzing data, but will also help reduce the overall testing time.

ELIGIBILITY:
Inclusion Criteria:

1. Able to communicate in either English or French
2. Impairment of central vision, affecting acuity due to any diagnosis
3. Visual acuity in the better eye with best standard correction of 20/60 or less
4. Potential benefit from magnification or other reading rehabilitation interventions, as determined by rehabilitation professional.
5. Client dossier with one of the partnering rehabilitation agencies.

Exclusion Criteria:

1. Complete blindness
2. Inability to communicate verbally
3. Inability to independently give informed written consent

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 38 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2023-03-28 (Actual); Study Completion 2023-03-28 (Actual)

PRIMARY OUTCOMES:
Rey Auditory Verbal Learning Test (RAVLT) | 15 minutes
  Participants are verbally presented with a list of 15 words that they are asked to repeat and memorize, then recall immediately, and again recall them 15 minutes later. The score is the number of items recalled from 0 to 15, with higher scores indicating better recall.
Letter Number Sequencing task | 2 minutes
  Participants are asked to speak out loud the first 13 letters of the alphabet and alternate them with consecutive numbers (e.g., 1 - A - 2 - B 3 -C ...). The score is the number of correct alternations between numbers and letter, from 0 to 26, with higher scores indicating better performance.
Montreal Cognitive Assessment - full or blind version | 4 minutes
  Participants are asked to complete the visual and auditory items of this cognitive screening measure. The Blind versions (no visual items is utilized for persons whose vision is too impaired to see the pictograms). The score is the total number of items completed correctly, ranging from 0 to 30 for the full version, and 0 to 22 for the Blind version, with higher scores indicating better outcomes
1-n-back task | 3 minutes
  Participants are asked to verbally repeat a string of numbers presented orally, while naming the previous item to the one just presented. The score is the total number of correct recalls, ranging from 0 to 25, with higher scores indicating better performance.

SECONDARY OUTCOMES:
Minnesota Reading Test (MNRead) | 2 minutes
  Participants are asked to read individual sentences on an eye chart. The log score indicates reading acuity ranging from -0.1 to 1.0 with higher numbers indicating poorer acuity.
Depression, Anxiety and Stress Scale | 5 minutes
  A 21-item questionnaire that measures the self-reported perception of depression, anxiety and stress on its three sub-scales, respectively. Scores for each item are from 0 to 3. Higher scores indicate higher levels of perceived depression, anxiety and stress, ranging each from 0 to 21 for each sub-scale.
Canadian Digit Triplet Test | 4 minutes
  A test measuring speech-in-noise perception. Participants are presented with three spoken digits through a head-set, and are asked to then enter them on a keyboard. Correct repetition will increase background noise, while incorrect answers will decrease background noise. The outcome measure is the estimated threshold for the signal-to-noise ratio where a participant can still comprehend the spoken digits. More negative score ratios indicate more tolerance to noise, therefore indicating better performance
Magnetic Resonance Imaging (MRI) - for subset of participants | 45 minutes
  Cortical invasive scan to measure structure and volume of brain regions involved in reading and sensory processing. Participants will placed in a Magnetic Resonance Imaging scanner in order to obtain structural measurement of their cortical architecture. Participants are asked to remain still a possible during these scans; however, they are not required to be otherwise engaged in any activity or decision-making. Higher volume measures indicate that more cortical volume is allocated to specific brain regions. This does not necessarily imply a functional judgment on its capacity, but is an anatomical measure only.

CONTACTS AND LOCATIONS:
Overall Officials: Walter Wittich, PhD, Principal Investigator — Université de Montréal
Locations (2):
- Canada (2):
  - Institut Nazareth et Louis-Braille du CISSS de la Montérégie-Centre, Longueuil, Quebec
  - Centre de réadaptation Lethbridge-Layton-Mackay du CIUSSS du Centre-Ouest-de-l'Île-de-Montréal, Montreal, Quebec

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wittich W, Pichora-Fuller MK, Johnson A, Joubert S, Kehayia E, Bachir V, Aubin G, Jaiswal A, Phillips N. Effect of Reading Rehabilitation for Age-Related Macular Degeneration on Cognitive Functioning: Protocol for a Nonrandomized Pre-Post Intervention Study. JMIR Res Protoc. 2021 Mar 11;10(3):e19931. doi: 10.2196/19931. PMID 33704074
- [Result] Aubin G, Phillips N, Jaiswal A, Johnson AP, Joubert S, Bachir V, Kehayia E, Wittich W. Visual and cognitive functioning among older adults with low vision before vision rehabilitation: A pilot study. Front Psychol. 2023 Mar 22;14:1058951. doi: 10.3389/fpsyg.2023.1058951. eCollection 2023. PMID 37034930
- See also: Open-access link for protocol publication — https://www.researchprotocols.org/2021/3/e19931

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2020-02-16): https://cdn.clinicaltrials.gov/large-docs/10/NCT04276610/Prot_SAP_000.pdf
  • Informed Consent Form (2020-02-07): https://cdn.clinicaltrials.gov/large-docs/10/NCT04276610/ICF_001.pdf